CLINICAL TRIAL: NCT03113786
Title: Efficacy of Amniotic Tissue (CLARIX 100 & CLARIX CORD 1K) in Pain Reduction and Improvement of Function in Low Back & Leg Pain in Discectomy Patients
Brief Title: CLARIX™ 100 & CLARIX CORD 1K for Discectomy Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amniox Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1001
Record Dates: First submitted 2017-04-06; First posted 2017-04-14 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Protruded Disk
Keywords: Discectomy; Lumbar discectomy; Protruding disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Subjects randomized to standard of care will undergo a traditional lumbar discectomy procedure without any additional interventions
- CLARIX™100 (Active Comparator): Subjects randomized to the CLARIX™100 arm will undergo a traditional lumbar discectomy, after which CLARIX™100 will be applied to the affected site. The tissue will be applied to the annulus at the defect site as a patch just prior to wound closure.
  Interventions: Other: CLARIX™100
- CLARIX CORD 1K (Active Comparator): Subjects randomized to the CLARIX CORD 1K arm will undergo a traditional lumbar discectomy, after which CLARIX CORD 1K will be applied to the affected site. The tissue will be applied to the annulus at the defect site as a patch just prior to wound closure.
  Interventions: Other: CLARIX CORD 1K

INTERVENTIONS:
Other: CLARIX™100 — CLARIX™100 is Amniox's processed and cryopreserved human amniotic membrane tissue retrieved from donated placental tissue after elective Cesarean Section delivery. Amniox's Amniotic Membrane is designated by the FDA as a tissue product under PHS 361 HCT/P (human cells, tissues and cellular and tissue-based products).
  Arms: CLARIX™100
Other: CLARIX CORD 1K — CLARIX CORD 1K is made from cryopreserved human umbilical cord, utilizing the patented CRYOTEK™ process. CLARIX CORD 1K is considered a Human Cells, Tissues & Cellular and Tissue-based product (HCT/P) by U.S. FDA standards.
  Arms: CLARIX CORD 1K

SUMMARY:
The purpose of the study is to evaluate the efficacy of CLARIX™ 100 and CLARIX™ CORD 1K as a tissue barrier when used as an annular patch in discectomy patients with low back & leg pain when compared to traditional discectomy patient outcomes. This will be a 120 patient, prospective randomized study model over a 5 year post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 90 years of age
* Patient is able to understand the aims and objectives of the trial and the trial procedures
* Patient is willing to give written informed consent to the trial
* Patient is able to follow up with regularly scheduled visits with and phone calls from Dr. Anderson and his research staff
* Diagnosed with lumbar protruding disc
* Suffer from radiating leg pain and low back pain that has failed a minimum of 6 months of conservative (non-operative) treatment options

Exclusion Criteria:

* Participation in clinical trial involving therapy for back pain within 30 days of screening
* Prior back surgery at the same level
* Inability to walk independently (adaptive devices such as walkers or canes are allowed)
* Relation (whether direct or indirect) to, student of, employee of, colleague of, indebted to the primary investigator, host institution or sponsoring company
* Receipt of corticosteroids, immunosuppressive agents, radiation therapy or chemotherapy within 1 month prior to visit
* Pregnancy or planning to become pregnant during study period
* Body Mass Index >50
* Patients with chronic diseases such as Crohn's disease, severe renal failure (serum creatinine 2.5 mg/dL or subject on hemodialysis), severe hepatic insufficiency: known cirrhosis, any degree of ascites, serum transaminases more than 3 times the upper limit of normal, life expectancy of less than one year, uncompensated or uncontrolled right sided heart failure with associated edema
* Severe anemia, hemoglobin <8.5 mg/dL
* Active, local or systemic malignancy such as lung cancer or leukemia
* Severe hypertension (systolic blood pressure greater than or equal to 200 mmHg or diastolic blood pressure greater than or equal to 100 mmHg)
* Severe hypoxia, with chronic oxygen or ventilation therapy
* History of collagen vascular disease or sickle cell anemia
* Active rheumatoid arthritis
* Systemic antibiotic therapy for any indication within 10 days of screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11-02 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Difference in low back & leg pain | 5 years
  To determine at various time points up to 5 years what, if any, difference there is between the three groups of 40 patients by using the Oswestry Disability Index scales for both back & leg pain
Difference in low back & leg pain | 5 years
  To determine at various time points up to 5 years what, if any, difference there is between the three groups of 40 patients by using the SF-12 scale for both back & leg pain
Difference in low back & leg pain | 5 years
  To determine at various time points up to 5 years what, if any, difference there is between the three groups of 40 patients by using the VAS for both back & leg pain

CONTACTS AND LOCATIONS:
Overall Officials: Scheffer Tseng, MD, PhD, Study Chair — BioTissue Holdings, Inc
Locations (1):
- Rothman Institute, Bensalem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No